CLINICAL TRIAL: NCT01412723
Title: EFICACIA DEL HIERRO AMINOQUELADO COMPARADO CON EL SULFATO FERROSO COMO COMPLEMENTO ALIMENTARIO EN PREESCOLARES CON DEFICIENCIA DE HIERRO.
Brief Title: Ferrous Sulfate Versus Iron Amino Acid Chelate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CES University (Other)
Collaborators: Nutreva S.A.S. (Unknown); Foundation Child Care - FAN (Other)
Responsible Party: Principal Investigator, Jose María Maya Mejía, Dean, CES University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SFHA-01
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Iron Deficiency
Keywords: Iron Deficiency; Child, Preschool; Dietary Iron; Ferrous sulfate; Bis-glycino iron II
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous sulphate (Active Comparator): Preschool children with depleted levels of iron enrolled in FAN Foundation of Medellin, which will be supplied with ferrous sulfate-fortified milk
  Interventions: Other: Ferrous sulfate as dietary supplementation
- Iron Amino acid chelate (Experimental): Preschool children with depleted levels of iron enrolled in FAN Foundation of Medellin , which will be supplied with iron amino acid chelate-fortified milk
  Interventions: Other: Iron amino acid chelated as dietary supplementation

INTERVENTIONS:
Other: Ferrous sulfate as dietary supplementation — Ferrous sulfate as dietary supplementation
  Arms: Ferrous sulphate
Other: Iron amino acid chelated as dietary supplementation — Iron amino acid chelated as dietary supplementation
  Arms: Iron Amino acid chelate

SUMMARY:
Iron deficiency and depleted levels of iron are the most prevalent nutritional deficiency and the leading cause of anemia in the world; this can occur at any age, but preschool children are at particular risk of developing it. This condition may cause serious repercussions for life, being a public health threat of considerable importance worldwide.

Food fortification is considered the most effective solution to counter this situation, because it can help more people than other solutions. It is going to carry out a community trial to compare the efficacy of ferrous sulfate with respect to iron amino acid chelate as a dietary supplement in preschool children of Medellin with depleted levels of iron; in terms of increasing ferritin levels in blood and maintain hemoglobin levels. It is hypothesized that at the end of the study the effect of milk fortified with iron amino acid chelate won't be less than the effect of fortified with ferrous sulfate.

It is hoped that the results may contribute, albeit indirectly, to improve the health status of children with depleted levels of iron whom consume iron-fortified products.

ELIGIBILITY:
Inclusion Criteria:

Children who

* Belong to institute FAN in Medellín
* Attend full time to institute FAN (eight hours)
* Have 2 to 5 years inclusive
* Submit depleted levels of iron (ferritin level equal to or less than 24 mg/L)

Exclusion Criteria:

Children who

* Submit anemia (hemoglobin level equal to or less than 11 g/dL)
* Have not stool analysis before intervention

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ferritin | Up to 8 weeks
  The Ferritin level in blood will be measured at the beginning of the study as one of the most important inclusion criteria. This also will be the base line of the study. After that randomization will be carried out and after two months (time frame which ferrous sulfate or iron aminoacid chelate would increase ferritin level in blood) ferritin level will be measured again as the primary outcome measure.

SECONDARY OUTCOMES:
Hemoglobin | Up to 8 weeks
  The Hemoglobin level in blood will be measured at the beginning of the study as one of the most important exclusion criteria. After that randomization will be carried out and after two months (time frame which ferrous sulfate or iron aminoacid chelate would increase ferritin level in blood) hemoglobin level will be measured again as one of secundary outcome measure. The hypothesis is that the hemoglobin level won't decrease
Infection | Daily. During 2 months of intervention
  Daily written report of the caregiver during the intervention
Adverse reaction | Daily. During 2 months of intervention
  The caregiver recorded daily if the child had an adverse reaction such as abdominal pain, nausea, vomiting, constipation, diarrhea, darkening of feces, and disgust for food.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Herrera, PhD en Patología, Study Director — CES University
Locations (1):
- Universidad CES, Medellín, Antioquia, Colombia